CLINICAL TRIAL: NCT05253040
Title: KEEP- A Randomised Feasibility Study of a Co-designed Physical Health Education Intervention to Improve Knowledge, Exercise Efficacy and Participation for Newly Diagnosed People With Parkinson's.
Brief Title: KEEP Intervention for People Newly Diagnosed With Parkinson's
Acronym: KEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Ledia Alushi, PhD Student, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A096150
Record Dates: First submitted 2022-02-02; First posted 2022-02-23 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: Physical activity; education; exercise; self-efficacy
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group will receive:
  Online education modules Online group discussions facilitated by Specialist Physiotherapist
  Interventions: Other: KEEP Intervention
- Control Group (Active Comparator): The comparator for this study is usual care pathway. Under the usual care pathway, participants will receive education booklets on exercise by Parkinson's UK.
  Interventions: Other: control

INTERVENTIONS:
Other: KEEP Intervention — Educational intervention
  Arms: Intervention group
Other: control — booklet from Parkinson's UK
  Arms: Control Group

SUMMARY:
Parkinson's Disease (PD) is a progressive neurological condition that affects movement, balance and cognition, resulting in loss of independence and compromised quality of life over the course of the condition. Research suggests that those detrimental outcomes can be reduced through physical activity (PA) and exercise, especially when those are started early. Educating people with Parkinson's (PwP) on the role of PA and exercise in PD progression can boost PA engagement by increasing enablers such as exercise self-efficacy and removing barriers such as misinformation about exercise and exercise outcomes.

Working closely with PwP and healthcare professionals, a physical health education programme was co-designed to address the needs and preferences of PwP around exercise and PA education. The process was supervised by the patient and Public Involvement group attended by PwP, academics, researchers and clinicians working with PwP.

The study will utilise an assessor blinded randomised controlled design to investigate the acceptability and feasibility of delivering an online physical health education programme for PwP who are newly diagnosed. Thirty PwP, diagnosed in the last 12-months, will be randomly allocated into two groups: 1) the intervention group in which participants will receive online education modules and will be invited to attend virtual group sessions with a specialist neuro-physiotherapist; 2) the control group which will follow the usual care pathway and participants will receive Parkinson's UK booklets.

The aim of the study is to explore an alternative approach to standard care regarding patient education in PD and evaluate the feasibility and acceptability of a co-designed education intervention for newly diagnosed PwP delivered online. Feasibility data will be collected during the study and acceptability data will be assessed via a questionnaire at the end. Outcomes including PA levels, exercise knowledge, exercise efficacy, and participation will be assessed at baseline, post-intervention and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Idiopathic Parkinson's Disease
* Within 12 months since diagnosis
* Stable medication regime for four weeks prior to initiation of trial
* Ability to understand written English

Exclusion Criteria:

* Acute illness
* History of neurological disorder other than Parkinson Disease
* Diagnosis of dementia or significant cognitive impairments
* Participation in NHS structured PD-specific education program with or without exercise classes in the last year
* Unable to understand written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2023-06-18 (Estimated)

PRIMARY OUTCOMES:
Acceptability assessment 1: Recruitment rate | Through study completion (12 months)
  Assessment of recruitment rate of study (% of eligible participants enrolled)
Acceptability assessment 2: Education programme compliance | Through study completion (12 months)
  Compliance with the online education programme (% of sessions completed)
Acceptability assessment 3: Drop out rate | Through study completion (12 months)
  Comparison of drop out rates (%) between the intervention group and control group
Acceptability assessment 4: Acceptability of Intervention | Completed at the end of participation in the study (after 8 weeks)
  A questionnaire designed to assess satisfaction with the education intervention. it includes multiple choice and open ended questions.
Feasibility of delivering the intervention online | Through study completion (12 months)
  Assessment of any technical problems or difficulties accessing online intervention as reported by participants

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale Part 3 | Baseline(week 0) and follow up (6-month post intervention)
  The UPDRS is the gold-standard scale for Parkinson's assessment and has four parts. For this study only UPDRS III, motor examination will be completed by a trained assessor. UPDRS III total scores range from 7 to 86 points, with higher scores indicating more severe impairment..
MiniBESTest | Baseline(week 0) and follow up (6-month post intervention)
  The Mini-BEST is a 14-item scale that assesses dynamic balance components including anticipatory postural adjustments, reactive postural control, sensory orientation and dynamic gait. The data is based on a total score of 28 points, with higher score indicating better task performance.
Five time Sit To Stand | Baseline(week 0) and follow up (6-month post intervention)
  Five time sit to stand is a validated test used to assess functional lower extremity strength, balance and risk falls in older adults. It has been used in PD population with high interrater and test-retest reliability. Longer time to complete indicates worse task performance.
Self-efficacy for Exercise | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  The Self-Efficacy for exercise (SEE) scale is a 9-item validated scale which assesses a person self-efficacy to exercise under different circumstances. This scale is a modified version of Bandura's Exercise Self-Efficacy Scale and ask participants to rate their perceived exercise efficacy on a scale form 0 meaning not confident at all to 10 meaning very confident. Higher score indicate higher self-efficacy
Hospital Anxiety and Depression Scale | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  Hospital Anxiety and Depression Scale (HADS) is a widely used questionnaire to measure anxiety and depression. A self-reported brief instrument which includes 14 questions aiming to detect and indicate severity of anxiety and depression. It has been used before and is a validated and reliable tool to use in Parkinson's population.
Apathy Evaluation Scale | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  Apathy Evaluation Scale (AES) is a standardised and validated self-rating instrument to evaluate apathy. It consists of 18 items that are scored on a 4-point Likert Scale, with highest score indicating more severe apathy
Multidimensional Outcome Expectation Scale | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  Outcome expectations about the benefits of regular exercise and PA will be measured by the Multidimensional Outcomes Expectations for Exercise Scale (MOEES). The MOEES has 15 items that reflect three subdomains of outcome expectations. The items were rated on a five-point scale from 1 (Strongly disagree) to 5 (Strongly agree) and summed to form the subscale measures of outcome expectations with higher scores reflecting greater beliefs about the benefits of regular exercise and physical activity.
Oxford Participation and Activities Questionnaire | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  Oxford Participation and Activities Questionnaire (Ox-PAQ) is a patient-reported outcome measure comprised of 23 items aiming to assess participation and activity in patients with long-term conditions.
Recent Physical Activity Questionnaire | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  Physical Activity will be measured subjectively and objectively. Subjectively it will be measured via the self-reported Recent Physical Activity Questionnaire (RPAQ), which is designed to assess PA in everyday life in the last 4 weeks. The questionnaire has three sections assessing a range of activities in different domains (around the house, work and recreation).
Knowledge of Exercise and Physical Activity | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  Knowledge of Exercise and Physical Activity questionnaire is a 10-item knowledge questionnaire around the role of exercise and physical activity in the management of PD and it has been designed by the PI to assess knowledge levels. A total score of 10 indicates better knowledge scores.
Wrist-worn accelerometer | Baseline(week 0), post intervention (week 8) and follow up (6-month post intervention)
  Objectively, physical activity will be measured with the use of a wrist-worn accelerometer (GeneActiv monitor) over 7 consecutive days.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Agley L, Hartley P, Duffill D, Iqbal A, Mackett A, Rennie KL, Lafortune L. Digital Intervention Promoting Physical Activity in People Newly Diagnosed with Parkinson's Disease: Feasibility and Acceptability of the Knowledge, Exercise-Efficacy and Participation (KEEP) Intervention. J Parkinsons Dis. 2024;14(6):1193-1210. doi: 10.3233/JPD-240071. PMID 39093079